CLINICAL TRIAL: NCT04660604
Title: Investigation of the Functional and Biomechanical Effect of Instrument Assisted Soft Tissue Mobilization Technique in Individuals With Asymptomatic Dynamic Knee Valgus - Randomized Controlled Trial
Brief Title: Investigation of the Effect of Instrument Assisted Soft Tissue Mobilization Technique in Individuals With Asymptomatic Dynamic Knee Valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IASTM-24.11.20
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Dynamic Knee Valgus; Force Production; Frontal Plan Projection Angle; Instrument-assisted Soft Tissue Mobilization; Postural Stability

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Masking Description: Participants do not have the knowledge about what we are investigated and group types.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Graston Technique® Group (Experimental): Participants were asked to warm up at a speed that they felt comfortable for 5 minutes at a gentle tempo with an ergometer. Time was followed by a stopwatch. Participants who completed warm-up were taken to GT® application. Application was implemented by a GT® certified therapist with 13 years of experience in orthopedic rehabilitation. Intervention dosage was determined as 2 times a week, 12 sessions over 6 weeks. GMed muscle was scanned between crista iliaca and trochanter major, and a fascial release was applied. Each session lasted 5 minutes. At the end of sessions, iliotibial band stretching exercises (30 seconds, 3 repetitions) was given to the treated side. Application protocol has been determined with reference to GT® manual
  Interventions: Device: Graston Technique®
- Control Group (No Intervention): Control group is followed up for 6 weeks without intervention.

INTERVENTIONS:
Device: Graston Technique® — Graston technique, one of the soft tissue mobilization techniques, has also been found to be effective method that affects muscle strength, performance and endurance through activation of muscle and nervous systems.
  Arms: Graston Technique® Group

SUMMARY:
STUDY DESIGN: Randomized controlled study OBJECTIVES: To investigate the contribution of instrument assisted soft tissue mobilization (IASTM) applied to gluteus medius (GMed) to isokinetic strength, femoral internal rotation (FIR), frontal plan projection angle (FPPA) and postural stability (PS) in individuals with asymptomatic dynamic knee valgus (DDV).

BACKGROUND: In the literature effect of IASTM on force production and performance has been examined with exercise, and results of the studies are contradictory. Studies investigating the effects of IASTM without exercise and at recommended dose are needed.

METHODS: 44 participants with DDV (21,39±1,79) were randomized to be control group (CG=22) and graston group (GG=22). First day, participants' FIR, FPPA with single leg squat test, dynamic and static PS on involved leg evaluations were completed. Second day, eccentric strength of GMed was measured by isokinetic test. IASTM application was applied 6 weeks, twice a week, 5 minutes, using Graston Technique® instruments. CG has not been attempted. Evaluations were repeated at the end of treatment.

DETAILED DESCRIPTION:
Introduction Dynamic knee valgus (DDV), one of the lower extremity faulty movement patterns, is a biomechanical deviation that occurs in 3 motion plans, involving femoral internal rotation (FIR) and contralateral pelvis fall simultaneously with hip adduction.1 Hip flexion, adduction and FIR moments occur simultaneously during loading phase of walking, running or landing after jumping. Combination of these moments also forms DDV. These moments are resisted by intrinsic moments caused by eccentric contractions of hip extensor, abductor and external rotator muscles. Strength deficiency of these muscles in weight transfer activities causes an increase in hip adduction, and FIR, changes whole lower extremity kinematics.2,3 The valgus alignment also increases the risk of injury.4 In the review examining relationship between hip muscle strength and DDV, it was determined that decrease in gluteus medius (GMed) strength in functional activities on single leg was associated with DDV.2 Abduction torque produced by hip abductors stabilizes pelvis on relatively fixed femur by controlling pelvis in frontal and horizontal planes during stance phase of walking and most of stance and GMed produces most of the compression forces in hip.3,5 Therefore, GMed strength is also very important for postural stability (PS). In individuals with DDV, strength of hip muscles, especially GMed, should be focused on increasing PS during the tests performed on single leg and in injury prevention programs.4,6 Anatomical features of women increase the risk of DDV. In addition, when gender comparison was made, it was seen that women needed more eccentric contraction in the hip abductor muscles during the stance phase of running.7, and strength deficiency in proximal hip stabilizers of females could cause a greater decrease in athletic performance compared to men.8 Therefore, evaluation of eccentric strength of GMed muscle should be evaluated specific to gender.2 Thus, a more precise conclusion can be found in terms of abductor muscle strength, DDV and lower extremity alignment.

Effect of soft tissue mobilization techniques on force production and performance is a remarkable topic. Instrument-assisted soft tissue mobilization (IASTM) technique, one of the soft tissue mobilization techniques, has also been found to be effective method that affects muscle strength, performance and endurance through activation of muscle and nervous systems.9-11 However, in studies IASTM technique was applied with an exercise protocol, and contribution of IASTM in force generation and performance increase is not understood.

According to our knowledge, in the literature there is no randomized controlled study examining the effect of IASTM applied without exercise. Aim of our study is to investigate changes caused by IASTM applied to GMed muscle on eccentric force production of GMed, FIR, frontal plane projection angle (FPPA) and PS.

ELIGIBILITY:
Inclusion Criteria:

* to be a female between ages of 18 and 35,
* to have an increase of more than 10 ° in FPPA in landing phase of single leg squat test (SLST),
* not to have pain complaints
* to be recreatively active.

Exclusion Criteria:

* body mass index of 30 kg/m² and above,
* to have previous lower extremity surgery and joint,
* meniscus or ligament injury,
* chronic knee instability,
* leg length inequality,
* joint degeneration detected by radiography,
* cardiac, musculoskeletal system, vestibular and neurological problems,
* using corticosteroids for a long time
* being pregnant.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — recreationally active, healthy females
Enrollment: 44 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in isokinetic strength measurement | Pre evaluation before the intervention, 1 day after the intervention
  gluteus medius eccentric strength evaluated with Cybex® Norm isokinetic dynamometer

SECONDARY OUTCOMES:
Change in postural stability evaluation | Pre evaluation before the intervention, 1 day after the intervention
  static and dynamic single leg postural stability
Change in Femoral internal rotation angle evaluation | Pre evaluation before the intervention, 1 day after the intervention
  Femoral internal rotation angle measurement
Change in frontal plan projection angle evaluation | Pre evaluation before the intervention, 1 day after the intervention
  Frontal plan projection angle measurement in single leg squat test

CONTACTS AND LOCATIONS:
Locations (1):
- Pelin Pişirici, Istanbul, Besiktas/Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided